CLINICAL TRIAL: NCT04927039
Title: Effects of Iloprost on Oxygenation During One-lung Ventilation in Supine-positioned Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2021-0465
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Mediastinal Mass
MeSH Terms: interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Drug: 5ml of inhaled normal saline
- Iloprost group (Experimental)
  Interventions: Drug: 20μg (2ml) of inhaled iloprost (Ventavis®) and 3ml of inhaled normal saline

INTERVENTIONS:
Drug: 5ml of inhaled normal saline — After the initiation of OLV, 5ml of normal saline is inhaled for 20 minutes using ultrasonic nebulizer, which is connected to the inspiratory limb of the ventilator system. Arterial blood gas analysis is performed 20 minutes after the completion of drug inhalation.
  Arms: Control group
Drug: 20μg (2ml) of inhaled iloprost (Ventavis®) and 3ml of inhaled normal saline — After the initiation of OLV, mixture of iloprost 2ml and normal saline 3ml is inhaled for 20 minutes using ultrasonic nebulizer, which is connected to the inspiratory limb of the ventilator system. Arterial blood gas analysis is performed 20 minutes after the completion of drug inhalation.
  Arms: Iloprost group

SUMMARY:
One-lung ventilation (OLV) is essential during mediastinal mass excision. However, OLV induces a drastic increase of intrapulmonary shunt due to maintained pulmonary perfusion through the nonventilated lung. In addition, it is reported that supine positioning of patient during OLV, which is required during mediastinal mass excision, results in worse oxygenation than lateral decubitus positioning.

Iloprost is a prostaglandin analogue and when inhaled during OLV, it acts selectively on the pulmonary vasculature, reducing pulmonary vascular resistance of well-ventilated lung and thereby alleviating ventilation-perfusion mismatch. The purpose of this study is to evaluate the effects of inhaled iloprost on oxygenation during one-lung ventilation in patients undergoing mediastinal mass excision.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for Video-assisted thoracoscopic surgery (VATS) mediastinal mass excision
2. Patient age from 20 to 80
3. American Society of Anaesthesiologists (ASA) physical status classification II~III

Exclusion Criteria:

1. Chronic obstructive pulmonary disease (COPD) with Forced expiratory volume in 1 second (FEV1) to Forced vital capacity (FVC) ratio < 0.7 and percentage of predicted FEV1 ≤ 80%
2. Diffusing capacity of carbon monoxide (DLCO) < 80%
3. Aspartate transaminase (AST) level ≥100 IU/mL or alanine transaminase (ALT) ≥ level 50 IU/L
4. Creatinine clearance ≤ 30mL/min
5. Congestive heart failure, arrhythmia
6. Unstable angina, coronary artery occlusive disease (CAOD), history of myocardial infarction within 6 months
7. Pulmonary edema, pulmonary arterial hypertension
8. Allergic to prostaglandin or prostacyclin analogue
9. Patients with peptic ulcer bleeding, trauma, intracranial hemorrhage
10. History of cerebrovascular disease (e.g. transient ischemic attack, stroke) within 3 months
11. Valvular heart disease
12. Pregnant women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-24 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
PaO2 (partial pressure of arterial oxygen) to FiO2 (fraction of inspired oxygen) ratio (P/F ratio) | Twenty minutes after the completion of drug inhalation
  The P/F ratio is a widely-used objective tool to identify hypoxemic respiratory failure when supplemental oxygen has been administered. It can be used to evaluate the effect of iloprost on oxygenation during OLV.

CONTACTS AND LOCATIONS:
Overall Officials: Kyuho Lee, Principal Investigator — Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No